CLINICAL TRIAL: NCT02672085
Title: In Vivo Clinical and Radiological Effects of Platelet-rich Plasma on Interstitial Supraspinatus Lesion: Randomized Study
Acronym: PRP Randomized
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Tour Hospital (Other)
Collaborators: Rive Droite SA (Unknown)
Responsible Party: Principal Investigator, Adrien Schwitzguebel, MD, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCPT PRP
Record Dates: First submitted 2015-06-05; First posted 2016-02-03 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Supraspinatis Interstitial Partial-thickness Tears; Platelet-rich Plasma (PRP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP infiltration (Experimental): Supraspinatus interstitial lesion needling and infiltration with PRP
  Interventions: Procedure: PRP infiltraiton
- Needling (Active Comparator): Supraspinatus interstitial lesion needling and infiltration with NaCl
  Interventions: Procedure: Needling

INTERVENTIONS:
Procedure: PRP infiltraiton — Two time with 1 month interval, PRP will be extracted from own blood's patients with Regenlab® extraction kit, and injected into supraspinatus interstitial lesion.
  Arms: PRP infiltration
Procedure: Needling — Two time with 1 month interval, saline water will be injected into supraspinatus interstitial lesion.
  Arms: Needling

SUMMARY:
Background and Rationale:

Tedious PRP infiltrations are emerging treatments for tendinopathies and tendon tears. It has been showed effective in different parts of the body, but current evidences for rotator cuff PRP infiltration remains poor. Some studies that tested infiltrations on transfixing lesions showed no statistically significant effect of PRP on tendon healing. The investigators believe that this might be explained by a "flushing effect" of PRP into subacromial space or glenohumeral joint. Therefore, it was decided to focus this study on interstitial lesions, in which PRP is entrapped into the lesion for a long time.

Objective:

The purpose of this study is to evaluate whether intra-tear PRP infiltrations promotes tear repair better than needling procedures of torn tendon in participants with supraspinatus interstitial tears.

As secondary objective, we will study symptoms alleviation in same way. Primary outcome: Primary outcome: Supraspinatus tear size change from baseline will be compared between cases receiving two PRP injections and controls receiving torn tendon needling, 6 months after second injection.

Secondary outcomes: Single Assessment Numeric Evaluation score, Constant score, ASES score, Shoulder pain disability index, and Visual analogue scale changes from baseline will be compared between cases receiving two PRP injections and controls receiving torn tendon needling, 0,1,3, and 6 months after second injection.

Study design: This case-control study is randomized 1:1 between PRP (intervention group) and needling (Control group). It is a superiority trial that will include 84 patients suffering from interstitial supraspinatus tears. As adjuvant therapy, patients from each arm will beneficiate from standard physical therapy program. PRP and needling will be repeated 2 times, at one month interval. First injection will occur up to two months after recruitment. Clinical follow-up will occur from second injection to one year after second injection, with clinical parameters evaluation at 0,1,3, and 6 months after second injection, and control MRI 6 months after second injection.

Study Product / Intervention: Supraspinatus tendon needling with intralesional PRP injection. PRP will be extracted with Regenlab® extraction kit. No other medications used.

Control Intervention (if applicable): Supraspinatus tendon needling with intralesional saline water injection.

Number of Participants with Rationale: 84 patients will be needed (37 in each group). A 10% of dropout has been taken in consideration.

Study Duration: 24 months from recruitment of the first patient to the last follow-up visit. Scientific report will be written within the two months following recruitment of the last patient.

Study Schedule: First-Participant-In: 01.6.2015 Last-Participant-Out: 30.6.2017

DETAILED DESCRIPTION:
DETAILLED PLANNED STATISTICAL METHODS

Hypothesis

Null hypothesis: In patients with interstitial rotator cuff tear, there is no difference in term of tendon tear size percentage between baseline and 6 months after intervention.

Alternative hypothesis: In patients with interstitial rotator cuff tear, there is a difference in term of tendon of tendon tear size percentage between baseline and 6 months after intervention.

Determination of Sample Size

No previous data allows predicting the standard deviation of supraspinatus tear volume. In order to evaluate the standard deviation of tear size progression in percentage from baseline, investigators aimed to identify patients followed conservatively for interstitial supraspinatus tears, and in which two MRI has been performed at 3 to 9 months of interval. In this way, 25 patients were identified, and their tear sizes were measured. From this sample, an hypothetical standard deviation of 76% of the initial teas size was estimated. The investigators considered that potential PRP effect on tear size is clinically relevant if it allows a healing of 50% of the lesion size. Taking on consideration those points, 76 patients should be included to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) of 80%. The Type I error probability associated with this test of this null hypothesis is 0.05. Taking in consideration 10% of potential dropouts, it was planned to include 84 patients.

Following planned Analyses will be performed by Dr Adrien Schwitzguébel at the end of the study:

* Baseline clinical parameters They will be compared between the two groups with adapted statistic tests (Chi-squared, Wilcoxon, or T test).
* Primary outcome Supraspinatus tear size percentage difference between baseline and 6 months post intervention will be compared between the two groups with Student test.
* Secondary outcome Clinical scores (Constant, ASES, SPADI, SANE, and VAS) differences between baseline and different time points will be compared between the two groups with Student test (or Wilcoxon test in case of non-parametric distribution). Even if those multiple analysis aims to evaluate clinical evolution of the two groups, no corrections will be applied on p values, but rather the aspect of a global tendency will be integrated in the discussion. In order to see whether small tears are more prone to beneficiate from treatment, correlation coefficient will be calculated between tear size percentage difference and initial tear size.
* Handling of missing data and drop-outs In case of missing clinical parameters on interest for primary outcome calculation, patients will be excluded of the study. In case of missing clinical parameters on interest for secondary outcome calculation or baseline clinical parameters, analysis will be performed by removing patients with the missing value from corresponding analysis only.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form),
* Symptomatic interstitial tear of the supraspinatus tendon,

Exclusion Criteria:

* Tear of infraspinatus or subscapularis tendons (same shoulder)
* Frozen shoulder (antepulsion deficit > 20%)
* Corticosteroid shoulder infiltration in the 3 months prior the inclusion,
* Patients suffering from symptomatic anaemia, or patients with severe cardiorespiratory insufficiency,
* Known or suspected non-compliance, drug or alcohol abuse,
* Patients incapable of judgement or under tutelage,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Lesion healing | 6 months
  After second PRP injection, tendon healing will be assessed by comparison of baseline MRI and control MRI

SECONDARY OUTCOMES:
Single Assessment Numeric Evaluation (SANE) score | 0,1,3, and 6 months, and last follow-up (12 months or more)
  Changes from baseline will be compared between cases receiving two PRP injections and controls receiving tendon needling, 0,1,3, and 6 months after second injection.
Pain Scores on the Visual Analogue Scale | 0,1,3, 6 months, and last follow-up (12 months or more)
  Changes from baseline will be compared between cases receiving two PRP injections and controls receiving tendon needling, 0,1,3, and 6 months after second injection.
Constant score | 0,1,3, and 6 months
  Changes from baseline will be compared between cases receiving two PRP injections and controls receiving tendon needling, 0,1,3, and 6 months after second injection.
ASES score | 0,1,3, and 6 months
  Changes from baseline will be compared between cases receiving two PRP injections and controls receiving tendon needling, 0,1,3, and 6 months after second injection.
Shoulder Pain Disability Index score | 0,1,3, and 6 months
  Changes from baseline will be compared between cases receiving two PRP injections and controls receiving tendon needling, 0,1,3, and 6 months after second injection.
Correlation between the initial tear size and the percentage of tear size evolution | 6 months
  The tear size change will be evaluated between the 2 MRI, at the baseline and at the 6 months endpoints. This correlation will be separately evaluated in each study arm, and in the whole sample.
Lesion healing between interstitial lesions that englobes or not the bone-tendon interface | 6 months
  Tendon healing will be assessed by comparison of baseline MRI and control MRI
Time limit in months from the first intervention to the last follow-up | 12-36 months
  Will be measurerd in months
Treatements at the end of the 6 months of PRP/Saline follow-up: Occurence of surgery | between 6 months and the last follow-up
  The occurence of surgery will be reported in both groups: cases receiving two PRP injections and controls
Treatements at the end of the 6 months of PRP/Saline follow-up: Occurence of corticoid infiltrations | between 6 months and the last follow-up
  The number of infiltrations of the subacromial with corticosteroids bursa will be reported in both groups: cases receiving two PRP injections and controls
Treatements at the end of the 6 months of PRP/Saline follow-up: Occurence of other infiltrations | between 6 months and the last follow-up
  The nature number of infiltrations of the subacromial bursa with others substances (i.e. PRP, sclerosing agents, autologous blood, hyaluronic acid, ...) will be reported in both groups: cases receiving two PRP injections and controls
Histological changes of tendon samples in case of surgery: tendon cellularity | between 6 months and the last follow-up
  Cells count will be compared between cases receiving two PRP injections and controls
Histological changes of tendon samples in case of surgery: vascularity | between 6 months and the last follow-up
  Vascularity (CD34+ blood vessels count) will be compared between cases receiving two PRP injections and controls
Histological changes of tendon samples in case of surgery: apoptosis | between 6 months and the last follow-up
  Apoptosis (p53+ cells count) will be compared between cases receiving two PRP injections and controls

CONTACTS AND LOCATIONS:
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwitzguebel AJ, Kolo FC, Tirefort J, Kourhani A, Nowak A, Gremeaux V, Saffarini M, Ladermann A. Efficacy of Platelet-Rich Plasma for the Treatment of Interstitial Supraspinatus Tears: A Double-Blinded, Randomized Controlled Trial. Am J Sports Med. 2019 Jul;47(8):1885-1892. doi: 10.1177/0363546519851097. Epub 2019 Jun 4. PMID 31161947